CLINICAL TRIAL: NCT05319197
Title: INVESTIGATION OF HAND FUNCTIONS IN CHILDREN WITH SPECIFIC LEARNING DISORDER
Brief Title: HAND FUNCTIONS OF CHILDREN WITH A SPECIFIC LEARNING DISORDER
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Other Study IDs: KutahyaHSUozgulogrenmeguclugu
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2022-04

CONDITIONS: Specific Learning Disability; Specific Learning Disorder; Fine Motor Skills; Hand Functions
MeSH Terms: conditions — Specific Learning Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SLD Group
  Interventions: Other: No Interventions
- Healthy Control Group
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — No Interventions

SUMMARY:
Children with Specific Learning Difficulties (SLD) may have problems with fine and gross motor skills compared to their healthy peers. These children may have poor manual dexterity. Taken together, it is not clear how motor and sensory competence of the hand are affected together. In this study, it was aimed to evaluate the sensory and motor ability of the hand and to compare the examined parameters between the SLD group and the healthy control group.

DETAILED DESCRIPTION:
Specific learning disability (SLD) is a common neurodevelopmental disorder that begins at school age and sometimes goes undetected until adulthood. Its incidence in school-aged children is about 5-15%. Children with SLD have difficulty in fulfilling academic qualifications. In addition, there are various problems with fine motor skills, motor-coordination, balance and gross motor skills.

Upper extremity speed and dexterity affect fine motor performance (as they involve manipulative tasks that require a certain amount of time and higher motor skills). In the literature, it is reported that manual dexterity is a stronger predictor than balance on the functional mobility of children with SLD, and it is emphasized that strategies to improve dexterity performance should be focused in interventions for fine motor skills for these children. In addition, it is demonstrated that taking the necessary precautions and planning by evaluating the gross and fine motor skills in detail in SLD is important for the independence and achievements of children in their daily living activities.

Weak hand skills are expected in children with SLD. Problems based on hand performance can be addressed in a more comprehensive way by comparing these children with children with typical development in terms of motor performance and functional mobility. Similarly, although it is recommended to evaluate senses such as touch and stereognosia when evaluating fine motor performance in these children, no comprehensive study including sensory and motor evaluations has been found in the literature.

In this study, in children with SLD; It is aimed to examine the limitations of hand motor and sensory functions in daily activities in terms of general motor competencies and hand skills of the child and to compare them with the healthy control group.

ELIGIBILITY:
Inclusion Criteria:

* To have a diagnosis of special learning disability (regarding DSM-V criteria)
* To be in the age range of 8-14

Exclusion Criteria:

* Any acute or chronic orthopedic or neurological disease that may affect walking performance,
* Any surgery within the last 6 months,
* Severe sensory (hearing, vision, etc.) impairment that prevents him/her from taking commands
* Cognitive and mental severe impairment

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Study Population: The convenience sampling will implement for this cross-sectional study. Children who have a diagnoisis of special learning disability regarding DSM-V criteria and who attends the Specific Learning Difficulty Support Education Program of the Ministry of National Education regularly twice a week will screen for eligibility by their physician and were subsequently requested to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Bruininks-Oseretsky Motor Proficiency Test- 2 Short Form (BOT-2SF) | 20 minutes
  Assesses fine motor precision, fine motor integration, and manual dexterity. Scores are reported as a percentile rank; higher scores indicate better fine motor skills.
Hand Grip Force | 10 minutes
  Changes from the baseline, To measure hand grip strength through Hydraulic Hand held Dynamo-meter. It will be measured in kilograms.
Pinch Grip Force | 6 minutes
  Participants were seated at a table on which the dynamometers were positioned. The subjects were told to keep their elbow flexed without resting their arm or the grip handle of the dynamometer on the table. Results will be evaluated in pounds.
Abilhand Kids | 5 minutes
  to assess for performance of activity. score range 0-42 point, higher scores mean a better outcome.
Minnesota Manual Dexterity Test | 25 minutes
  to assess manual dexterity, higher scores mean a worse outcome.
Sensory Function | 30 minutes
  Proprioception, stereognosis, and two-point discrimination will be tested. Lower scores indicate better sensory function.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail SARAÇOĞLU, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Afyonkarahisar Özel Eğitim ve Rehabilitasyon Merkezi, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No